CLINICAL TRIAL: NCT07123142
Title: Evaluation of Steroidogenesis Disorders in Patients With Friedreich's Ataxia: A Clinical Pilot Study
Brief Title: FRIEDREICH ATAXIA- STEROIDOGENESIS
Acronym: FRIEDSTERO
Status: Recruiting | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Ozge Bayrak Demirel, MD, Pediatric Endocrinologist, Istanbul University
Other Study IDs: ITF_FERREDOX; CEDD2025_FAS_Study (Other: Çocuk Endokrin ve Diyabet Derneği)
Record Dates: First submitted 2025-08-08; First posted 2025-08-14 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Friedreich's Ataxia; Steroidogenesis
Keywords: Friedreich's ataxia; steroidogenesis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Friedreich's ataxia group: Genetically confirmed FA
- Healthy Control Group: not having any known disease and being similar age, sex and pubertal status with the disease group

SUMMARY:
Friedreich's ataxia (FA) is a rare autosomal recessive disorder caused by GAA repeat expansion in the FXN gene, leading to impaired iron-sulfur (Fe-S) cluster biosynthesis and mitochondrial dysfunction. Fe-S clusters are essential for the function of several enzymes involved in steroid hormone production. While animal and cell culture studies suggest impaired steroidogenesis in FA, no clinical study has systematically evaluated this in human patients. This pilot study aims to investigate adrenal and gonadal steroidogenesis pathways in FA patients using LC-MS/MS-based steroid profiling. A total of 11 genetically confirmed FA patients followed at Istanbul Faculty of Medicine will be enrolled. Clinical data and serum samples will be collected and compared with those of 15 age- and sex-matched healthy controls. The findings are expected to enhance understanding of endocrine alterations in FA and guide future therapeutic approaches.

DETAILED DESCRIPTION:
Friedreich's ataxia (FA) is characterized by mitochondrial dysfunction due to impaired iron-sulfur (Fe-S) cluster formation caused by GAA repeat expansion in the FXN gene. Fe-S clusters are crucial for the activity of several mitochondrial enzymes, including cytochrome P450 family members such as CYP11A1, CYP11B1, and CYP11B2, which are involved in the biosynthesis of steroid hormones. These enzymes require ferredoxin and ferredoxin reductase, whose function also depends on Fe-S clusters. Experimental studies have shown reduced levels of testosterone and progesterone in FA models, suggesting that steroidogenesis is disrupted in FA. This study will evaluate the steroid profiles of FA patients via LC-MS/MS, compare them with healthy controls, and investigate correlations with age, sex, and disease severity. It will be the first clinical study to address steroidogenic defects in FA patients.

ELIGIBILITY:
Inclusion Criteria (FA Group):

* Genetically confirmed Friedreich's Ataxia diagnosis
* Signed informed consent (parents and/or participants depending on age)

Inclusion Criteria (Control Group):

* Healthy individuals with no known chronic or endocrine disease
* Age- and sex-matched to FA patients
* Signed informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study includes patients diagnosed with Friedreich's ataxia (FRDA) aged 7 to 33 years and age- and sex-matched healthy controls. All participants are followed in pediatric and adult endocrinology outpatient clinics. The study group consists of 11 FRDA patients (3 females, 8 males), and the control group consists of 15 healthy individuals (5 females, 10 males). Both prepubertal and pubertal subjects are included.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Serum steroid hormone and intermediate metabolite levels | 3 months
  Serum steroid hormone and intermediate metabolite levels (e.g., progesterone, testosterone, DHEA, cortisol, etc.) measured via LC-MS/MS (Time Frame: within 1 month of sampling)

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The study involves sensitive individual patient data collected in a clinical setting. Due to ethical concerns, data privacy regulations, and the limited sample size that may risk re-identification, individual participant data (IPD) will not be shared.

REFERENCES:
- [Background] Zhang S, Napierala M, Napierala JS. Therapeutic Prospects for Friedreich's Ataxia. Trends Pharmacol Sci. 2019 Apr;40(4):229-233. doi: 10.1016/j.tips.2019.02.001. PMID 30905359